CLINICAL TRIAL: NCT02745795
Title: Motivational Intervention Through the Generation of an Interpersonal Plan About Nutrition and Physical Exercise Study (IMAGINE Study), a Randomized Controlled Trial With Obese and Overweight Adolescents in Portuguese High Schools
Brief Title: Efficacy of Motivational Interview in the Treatment of Obesity and Overweight in Adolescents
Acronym: IMAGINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro Hospitalar Lisboa Norte (Other)
Collaborators: University of Lisbon (Other); Faculdade de Psicologia e de Ciências de Educação da Universidade do Porto (Unknown)
Responsible Party: Principal Investigator, Maria do Céu Machad, Director of the Department of Pediatry of Centro Hospitalar Lisboa Norte, Chair of Pediatry at Medicine School of the University of Lisbon, Centro Hospitalar Lisboa Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CC-336
Record Dates: First submitted 2016-04-05; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Obesity
Keywords: Motivational interview; adolescents; obesity; overweight; physical activity; diet
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MIG: Motivational Interview Group (Experimental): Group submitted to three face-to-face interviews using motivational interview techniques to elicit motivation for adhesion to a diet and physical activity plan intended to loose weight. The interviews will be done at schools with three months intervals.
  Interventions: Behavioral: Motivational Interview
- CIG: Conventional Intervention Group (Sham Comparator): Group submitted to three face-to-face interviews without using motivational interview techniques to elicit motivation for adhesion to a diet and physical activity plan intended to loose weight. The interviews will be done at schools with three months intervals.
  Interventions: Behavioral: Conventional Interview

INTERVENTIONS:
Behavioral: Motivational Interview — Three face-to-face interviews using motivational interview techniques to elicit motivation for adhesion to a diet and physical activity plan intended to loose weight. The interviews will be done at schools with three months intervals.
  Arms: MIG: Motivational Interview Group
Behavioral: Conventional Interview — Three face-to-face interviews without using motivational interview techniques to elicit motivation for adhesion to a diet and physical activity plan intended to loose weight. The interviews will be done at schools with three months intervals.
  Arms: CIG: Conventional Intervention Group

SUMMARY:
The objective of the study is to investigate the efficacy of motivational interview intervention with adolescent students at a school environment on the adhesion to a therapeutic plan to loose weight.

DETAILED DESCRIPTION:
Motivational interview (MI) is a style of communication collaborative, objective-directed, with special attention to change talk.

The present study's main objective is to investigate the efficacy of a MI intervention in adolescents with weight excess, in a school setting, over their motivation to adhere to a health lifestyle plan of dietary habits and physical exercise.

Secondary objectives are to investigate the effect of MI over self-concept, quality of life, depressive symptoms, anxiety symptoms, body mass index, abdominal circumference and blood pressure.

Registry Procedures Data on anthropometric parameters is recorded in data collection sheet and stored in individual files, which are available for monitoring procedures and for auditing by the Metabolic and Food Behavior Disorders Scientific Committee.

Data Checks Data checks will be performed to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry

Source Data Verification All the data will be checked to assess accuracy, completeness, or representativeness of registry data by comparing the data to external data sources: audio-taped interviews, paper case report forms and paper case self-report forms. All the registries will be stored during five years after study completions according to the Medical Faculty of Lisbon norms.

Variables:

Motivational Interview Audio-taped clinical interview record Motivational Interviewing Treatment Integrity (MITI) version 3.1.1

Motivation to adhere to a physical exercise plan Self-report by a paper questionnaire Self-regulation and perceived competence questionnaire to begin or maintain an healthy diet

Motivation to adhere to a diet plan Self-report by a paper questionnaire Self-regulation and perceived competence questionnaire to begin or maintain regular physical exercise

Self-concept Self-report by a paper questionnaire Self Perception Profile for Children

Quality of life Self-report by a paper questionnaire Pediatric Quality of Life Inventory 4.0 (PEDSQL 4.0)

Depressive symptoms Self-report by a paper questionnaire Children Depression Inventory (CDI)

Anxiety symptoms Self-report by a paper questionnaire State-Trait Anxiety Inventory for Children (STAIC C-2)

Body mass index Calculated by the ratio of weight in kilograms over the square of height in meters^2.

Weight Direct measurement by the research team Measured with Omron Body Composition Monitor with Scale BF 11® (Omron®, Kyoto, Japan) in kilograms

Height Direct measurement by the research team Measured with Seca® 213 Portable Stadiometer Height-Rod® (Seca@, Hamburg, Germany) in meters

Abdominal circumference Direct measurement by the research team Seca 203 Circumference Measuring Tape® (Seca@, Hamburg, Germany) in centimeters

Blood pressure Direct measurement by the research team Riester Risan Sphygmomanometer® (Riester®, Jungingen, Germany) in mm Hg

ELIGIBILITY:
Inclusion Criteria:

* Age between 14 and 19 years old
* Body mass index percentile equal or above 85th percentile according to World Health Organization charts (de Onis 2010)

Exclusion Criteria (one or more of the following):

* recent weight loss of 10% or more of body weight
* pregnancy
* breastfeeding
* endocrine disease
* present therapy with antidepressant or hypoglycemic drugs
* present treatment for food behavior disease or depression
* cognitive impairment of the student or his/her legal tutor.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Motivation scores to adhere to a diet and physical activity plan | Six months
  Motivation scores assessed by two self-report confidential paper questionnaires (Self-regulation and perceived competence questionnaire to begin or maintain an healthy diet and Self-regulation and perceived competence questionnaire to begin or maintain regular physical exercise)

SECONDARY OUTCOMES:
Self-concept score | Six months
  Self-report score assessed by a paper questionnaire (Self Perception Profile for Children)
Quality of life score | Six months
  Quality of life score assessed by Pediatric Quality of Life Inventory 4.0 (PEDSQL 4.0)
Depressive symptoms score | Six months
  Depressive symptoms score assessed by Children Depression Inventory (CDI)
Anxiety symptoms | Six months
  Anxiety score symptoms assessed by State-Trait Anxiety Inventory for Children (STAIC C-2)
Abdominal circumference in centimeters | Six months
  Abdominal circumference measured with Seca 203 Circumference Measuring Tape® (Seca@, Hamburg, Germany)
Blood pressure in mm Hg | Six months
  Blood pressure measured with Riester Risan Sphygmomanometer® (Riester®, Jungingen, Germany)
Weight in kilograms | Six months
  Weight measured with Omron Body Composition Monitor with Scale BF 11® (Omron®, Kyoto, Japan)
Height in meters | Six months
  Height in meters measured with Seca® 213 Portable Stadiometer Height-Rod® (Seca@, Hamburg, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Serra-de-Lemos, PhD, Study Chair — Faculty of Psychology and Education Sciences of University of Porto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Physical Activity Guidelines Advisory Committee report, 2008. To the Secretary of Health and Human Services. Part A: executive summary. Nutr Rev. 2009 Feb;67(2):114-20. doi: 10.1111/j.1753-4887.2008.00136.x. No abstract available. PMID 19178654
- [Background] Hettema J, Steele J, Miller WR. Motivational interviewing. Annu Rev Clin Psychol. 2005;1:91-111. doi: 10.1146/annurev.clinpsy.1.102803.143833. PMID 17716083
- [Background] Bean MK, Mazzeo SE, Stern M, Bowen D, Ingersoll K. A values-based Motivational Interviewing (MI) intervention for pediatric obesity: study design and methods for MI Values. Contemp Clin Trials. 2011 Sep;32(5):667-74. doi: 10.1016/j.cct.2011.04.010. Epub 2011 Apr 29. PMID 21554994
- [Background] Tanofsky-Kraff M, Shomaker LB, Wilfley DE, Young JF, Sbrocco T, Stephens M, Ranzenhofer LM, Elliott C, Brady S, Radin RM, Vannucci A, Bryant EJ, Osborn R, Berger SS, Olsen C, Kozlosky M, Reynolds JC, Yanovski JA. Targeted prevention of excess weight gain and eating disorders in high-risk adolescent girls: a randomized controlled trial. Am J Clin Nutr. 2014 Oct;100(4):1010-8. doi: 10.3945/ajcn.114.092536. Epub 2014 Aug 13. PMID 25240070
- [Background] de Onis M, Lobstein T. Defining obesity risk status in the general childhood population: which cut-offs should we use? Int J Pediatr Obes. 2010 Dec;5(6):458-60. doi: 10.3109/17477161003615583. Epub 2010 Mar 17. No abstract available. PMID 20233144
- [Background] Aviram A, Westra HA. The impact of motivational interviewing on resistance in cognitive behavioural therapy for generalized anxiety disorder. Psychother Res. 2011 Nov;21(6):698-708. doi: 10.1080/10503307.2011.610832. Epub 2011 Aug 31. PMID 21878034
- [Background] Kosti RI, Panagiotakos DB. The epidemic of obesity in children and adolescents in the world. Cent Eur J Public Health. 2006 Dec;14(4):151-9. doi: 10.21101/cejph.a3398. PMID 17243492
- [Background] Resnicow K, Jackson A, Wang T, De AK, McCarty F, Dudley WN, Baranowski T. A motivational interviewing intervention to increase fruit and vegetable intake through Black churches: results of the Eat for Life trial. Am J Public Health. 2001 Oct;91(10):1686-93. doi: 10.2105/ajph.91.10.1686. PMID 11574336
- [Background] Faria L. Harter's self-perception profile for children adapted for use with young Portuguese students. Percept Mot Skills. 2001 Jun;92(3 Pt 1):711-20. doi: 10.2466/pms.2001.92.3.711. PMID 11453198
- [Background] Gee S, Chin D, Ackerson L, Woo D, Howell A. Prevalence of childhood and adolescent overweight and obesity from 2003 to 2010 in an integrated health care delivery system. J Obes. 2013;2013:417907. doi: 10.1155/2013/417907. Epub 2013 Jul 18. PMID 23970960
- [Background] Kovacs M. The Children's Depression, Inventory (CDI). Psychopharmacol Bull. 1985;21(4):995-8. No abstract available. PMID 4089116
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Gidding SS, Dennison BA, Birch LL, Daniels SR, Gillman MW, Lichtenstein AH, Rattay KT, Steinberger J, Stettler N, Van Horn L; American Heart Association; American Academy of Pediatrics. Dietary recommendations for children and adolescents: a guide for practitioners: consensus statement from the American Heart Association. Circulation. 2005 Sep 27;112(13):2061-75. doi: 10.1161/CIRCULATIONAHA.105.169251. PMID 16186441
- [Background] Neumark-Sztainer DR, Friend SE, Flattum CF, Hannan PJ, Story MT, Bauer KW, Feldman SB, Petrich CA. New moves-preventing weight-related problems in adolescent girls a group-randomized study. Am J Prev Med. 2010 Nov;39(5):421-32. doi: 10.1016/j.amepre.2010.07.017. PMID 20965379
- [Background] Flattum C, Friend S, Story M, Neumark-Sztainer D. Evaluation of an individualized counseling approach as part of a multicomponent school-based program to prevent weight-related problems among adolescent girls. J Am Diet Assoc. 2011 Aug;111(8):1218-23. doi: 10.1016/j.jada.2011.05.008. PMID 21802570
- [Background] Feinson J, Atkinson A, Hassink S. How a primary care quality improvement initiative is implementing the expert recommendations on childhood obesity. Del Med J. 2010 Feb;82(2):57-65. PMID 20369454
- [Background] Lang PJ, Bradley MM. Emotion and the motivational brain. Biol Psychol. 2010 Jul;84(3):437-50. doi: 10.1016/j.biopsycho.2009.10.007. Epub 2009 Oct 30. PMID 19879918
- [Background] Wang Y, Lobstein T. Worldwide trends in childhood overweight and obesity. Int J Pediatr Obes. 2006;1(1):11-25. doi: 10.1080/17477160600586747. PMID 17902211
- [Background] Resnicow K, Davis R, Rollnick S. Motivational interviewing for pediatric obesity: Conceptual issues and evidence review. J Am Diet Assoc. 2006 Dec;106(12):2024-33. doi: 10.1016/j.jada.2006.09.015. PMID 17126634
- [Background] Neumark-Sztainer D, Story M, Hannan PJ, Rex J. New Moves: a school-based obesity prevention program for adolescent girls. Prev Med. 2003 Jul;37(1):41-51. doi: 10.1016/s0091-7435(03)00057-4. PMID 12799128
- [Background] Ryan RM, Deci EL. Intrinsic and Extrinsic Motivations: Classic Definitions and New Directions. Contemp Educ Psychol. 2000 Jan;25(1):54-67. doi: 10.1006/ceps.1999.1020. PMID 10620381
- [Background] Ball GD, Mackenzie-Rife KA, Newton MS, Alloway CA, Slack JM, Plotnikoff RC, Goran MI. One-on-one lifestyle coaching for managing adolescent obesity: Findings from a pilot, randomized controlled trial in a real-world, clinical setting. Paediatr Child Health. 2011 Jun;16(6):345-50. doi: 10.1093/pch/16.6.345. PMID 22654546
- [Background] Flattum C, Friend S, Neumark-Sztainer D, Story M. Motivational interviewing as a component of a school-based obesity prevention program for adolescent girls. J Am Diet Assoc. 2009 Jan;109(1):91-4. doi: 10.1016/j.jada.2008.10.003. PMID 19103327
- [Background] Burke BL, Arkowitz H, Menchola M. The efficacy of motivational interviewing: a meta-analysis of controlled clinical trials. J Consult Clin Psychol. 2003 Oct;71(5):843-61. doi: 10.1037/0022-006X.71.5.843. PMID 14516234
- [Background] Council on Sports Medicine and Fitness; Council on School Health. Active healthy living: prevention of childhood obesity through increased physical activity. Pediatrics. 2006 May;117(5):1834-42. doi: 10.1542/peds.2006-0472. PMID 16651347
- [Background] Moyers TB, Martin T, Manuel JK, Hendrickson SM, Miller WR. Assessing competence in the use of motivational interviewing. J Subst Abuse Treat. 2005 Jan;28(1):19-26. doi: 10.1016/j.jsat.2004.11.001. PMID 15723728
- [Background] Lurbe E, Cifkova R, Cruickshank JK, Dillon MJ, Ferreira I, Invitti C, Kuznetsova T, Laurent S, Mancia G, Morales-Olivas F, Rascher W, Redon J, Schaefer F, Seeman T, Stergiou G, Wuhl E, Zanchetti A; European Society of Hypertension. Management of high blood pressure in children and adolescents: recommendations of the European Society of Hypertension. J Hypertens. 2009 Sep;27(9):1719-42. doi: 10.1097/HJH.0b013e32832f4f6b. PMID 19625970
- [Background] Irby M, Kaplan S, Garner-Edwards D, Kolbash S, Skelton JA. Motivational interviewing in a family-based pediatric obesity program: a case study. Fam Syst Health. 2010 Sep;28(3):236-46. doi: 10.1037/a0020101. PMID 20939628
- [Background] National High Blood Pressure Education Program Working Group on High Blood Pressure in Children and Adolescents. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. Pediatrics. 2004 Aug;114(2 Suppl 4th Report):555-76. No abstract available. PMID 15286277
- [Derived] Freira S, Lemos MS, Fonseca H, Williams G, Ribeiro M, Pena F, do Ceu Machado M. Anthropometric outcomes of a motivational interviewing school-based randomized trial involving adolescents with overweight. Eur J Pediatr. 2018 Jul;177(7):1121-1130. doi: 10.1007/s00431-018-3158-2. Epub 2018 May 15. PMID 29766325